CLINICAL TRIAL: NCT04297228
Title: Step by Step: A Family-Centered Healthy Lifestyle Intervention
Brief Title: Pediatric Obesity Treatment in a Safety Net Clinic: Piloting the Step by Step Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Community Volunteers In Medicine (Other)
Collaborators: American Academy of Pediatrics (Other)
Responsible Party: Principal Investigator, Kimberly Stone, Pediatrician, Community Volunteers In Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20560
Record Dates: First submitted 2020-02-25; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Pediatric Obesity; Overweight and Obesity
Keywords: pediatric obesity; safety net clinic; patient centered; nutrition therapy; body weight
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity; Body Weight

STUDY DESIGN:
Intervention Model Description: Pilot Program to Implement a Family Centered Pediatric Obesity Treatment Program in a Safety Net Clinic using Goal Setting Principles and Behavior Change Theory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Step by Step Program (Experimental): Thirteen 1.5 hour weekday educational sessions, five 1-hour weekday fitness classes and seventeen 1 hour weekend walks/farmer's market trips were scheduled over 22 weeks. The planned total contact time was 41.5 hours, above the minimum effective amount and recommended by the USPSTF. Children participated in all activities. Weekly text messages with motivational messages and reminders were planned.
  Educational Topics included:
  Intro and Goal Setting How to Read Nutrition Labels How to Build a Healthy Meal Choose My Plate/Walking for Fitness Healthy Fast Food Add More Fruits/Vegetables to Meals Add More Physical Activity Each Day Healthy Snacks and Drinks Healthy Desserts Circuit Training at Home Favorite Recipe Makeover Step by Step Jeopardy Celebration of Completion
  Interventions: Behavioral: Step by Step: A Family-Centered Healthy Lifestyle Intervention

INTERVENTIONS:
Behavioral: Step by Step: A Family-Centered Healthy Lifestyle Intervention

SUMMARY:
Obesity treatment interventions have been studied in pediatric primary care offices and are often conducted in low-income and minority populations, and pediatric obesity clinics. Key components of programs that have been shown to be effective include parent engagement providing physical activity, nutrition and behavior education and at least 26 hours of total contact time. However, there is little guidance in the literature describing translation of successful programs into sustainable, real-world practice for uninsured children and families. To the investigator's knowledge no studies in the United States have evaluated the feasibility of implementing a fitness and nutrition program in safety net clinics where uninsured parents and their children receive health care. The objectives of this project were to design an evidence-based, family-centered fitness and nutrition program and evaluate the feasibility and acceptability of implementing this program in a Volunteer in Medicine Clinic, discussing successes, challenges and lessons learned.

DETAILED DESCRIPTION:
The objectives of this project were to design an evidence-based, family-centered fitness and nutrition program and evaluate the feasibility and acceptability of implementing this program in a Volunteer in Medicine Clinic, discussing successes, challenges and lessons learned.

This prospective pilot study was conducted within a Volunteers in Medicine (VIM) model clinic in Southeastern Pennsylvania from July - December 2012. The VIM Model focuses on providing primary care to children, adolescents and adults that are uninsured. This model is guided by the principles of inclusion, service and community involvement, with volunteers providing the vast majority of health care and support services.

Community Volunteers in Medicine (CVIM) provides primary care and dental care to uninsured adults and children who live or work in Chester County with incomes less than 300% of the federal poverty level. In 2016, Chester County's residents were 7% Hispanic, 24% obese, 9% uninsured and 10% of children living in families with incomes below the poverty level. Most pediatric patients served by CVIM are of Hispanic/Latino descent and have a high prevalence of overweight and obesity (54%), which is higher than the county prevalence of 25% in school-aged children.

After a quality improvement project identified the high prevalence of childhood obesity in children served by CVIM, the authors proposed developing a family-centered obesity treatment program. CVIM's Executive Board committed support to the program. Temple University School of Medicine's Institutional Review Board approved the project. Consent materials were available in English and Spanish.

The program name Step by Step (Paso a Paso) was chosen by consensus, logo designed by a local graphic artist, and T-shirts provided to staff, volunteers and participants. Behavior change theory and goal-setting principles informed the program design. A literature review identified evidence-based best practices. Thirteen 1.5 hour weekday educational sessions, five 1-hour weekday fitness classes and seventeen 1 hour weekend activities were scheduled over 22 weeks. The planned total contact time was 41.5 hours, above the minimum effective amount recommended by the USPSTF. Children participated in all activities. Weekly text messages with motivational messages and reminders were planned. A Manual of Operations detailed the volunteer orientation, session outlines, and handouts. Sessions had bilingual staff and handouts were available in English and in Spanish. Clinic staff, volunteers and family members were encouraged to participate in fitness and nutrition activities.

Staff and Volunteer Recruitment and Training Providers recruited from clinic volunteers and staff conducted enrollment histories and physical examinations. The clinic's nutrition education specialist organized cooking classes with assistance from volunteers. Volunteers recruited from an Accelerated Pre-Medicine Post Bachelor's Program at a local college completed a background check, CVIM volunteer orientation and Step by Step program orientation. Volunteers provided child supervision, assistance with physical activity and cooking classes and language support. A physician (KS) was present for every session.

Participant Recruitment and Enrollment Enrollment goal was 10 families. Chart review identified eligible families; they were contacted by phone and invited to attend the enrollment meeting with a standard script.

At enrollment, parents signed informed consent and children assented; parents gave permission for photography and physical activity participation. Parents and children completed baseline questionnaires on fitness and nutrition knowledge and practices. Participant histories and physicals were completed using the Pennsylvania Sports Physical Standard form. Families gave permission to receive text reminders and were given a schedule for activities and educational sessions.

ELIGIBILITY:
Inclusion Criteria:

* Families were eligible if at least one parent and one child received healthcare at CVIM with a BMI of >75%ile for age

Exclusion Criteria:

* none

Ages: 4 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06-12 (Actual); Primary Completion 2012-12-17 (Actual); Study Completion 2012-12-17 (Actual)

PRIMARY OUTCOMES:
Attendance at Sessions | 22 weeks
  Numerator: Number of Families attending/Denominator: Number of sessions Numerator: Number of Fathers AttendingDenominator: Number of Sessions Numerator: Number of Children attending/Denominator: Number of sessions.

SECONDARY OUTCOMES:
BMI | 22 weeks
  Pre and Post Intervention BMI measurements on all family

IPD SHARING:
Plan to Share IPD: No
We are not sharing any individual participant data

REFERENCES:
- See also: Community Volunteers in Medicine website — http://www.cvim.org